CLINICAL TRIAL: NCT01459003
Title: Evaluation of Beauty Care Before Chemotherapy in Women With Breast Cancer
Acronym: BEAUTY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2011-A00811-40; 2010/1632 (Other: CSET number)
Record Dates: First submitted 2011-10-24; First posted 2011-10-25 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

ARMS (2):
- experimental (Experimental)
  Interventions: Other: beauty care
- control (No Intervention)

INTERVENTIONS:
Other: beauty care — beauty care performed before each chemo cycle
  Arms: experimental

SUMMARY:
Evaluation of beauty care in women receiving adjuvant chemotherapy for breast cancer

ELIGIBILITY:
Inclusion Criteria:

* breast cancer with no metastasis receiving adjuvant chemotherapy

Exclusion Criteria:

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
quality of life questionnaire | up to 12 months
  body image

CONTACTS AND LOCATIONS:
Overall Officials: Mahasti Saghatchian, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, Val de Marne, France

REFERENCES:
- [Derived] Saghatchian M, Lacas B, Charles C, Ghouadni A, Clain GT, Boinon D, Delaloge S, Vaz-Luis I, Dauchy S, Amiel P. BEAUTY and the breast: is adjuvant chemotherapy the right time for a beauty boost? Lessons learned from a large randomized controlled trial. Qual Life Res. 2022 Mar;31(3):723-732. doi: 10.1007/s11136-021-02947-6. Epub 2021 Jul 29. PMID 34324138